CLINICAL TRIAL: NCT03182829
Title: Post Marketing Study of an in Vitro Diagnostic Test for Direct Oral Anticoagulants (Apixaban, Edoxaban, Rivaroxaban, Dabigatran) in Urine
Brief Title: In Vitro Diagnostic Test for DOAC in Urine
Acronym: PADOASU
Status: Completed | Type: Observational
Sponsor: Doasense GmbH (Industry)
Collaborators: CRS Clinical Research Services Mannheim GmbH (Industry); Heidelberg University (Other); Medical Care Center Dr. Limbach and Colleagues, Heidelberg, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: DOA-CS-002
Record Dates: First submitted 2017-06-08; First posted 2017-06-09 (Actual); Results first posted 2021-05-04 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-03

CONDITIONS: Anticoagulant Therapy
Keywords: direct oral anticoagulants; apixaban; dabigatran; edoxaban; rivaroxaban; urine; LC-MS/MS; evaluation study; point of care test; blood coagulation; coagulation test; anticoagulant; thrombosis; pulmonary embolism; atrial fibrillation; anticoagulation; mass spectrometry; POC test
MeSH Terms: conditions — Thrombosis; Pulmonary Embolism; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine sample, spontaneously collected from patients
  "publication Thromb Haemost. 2019 Nov 8. doi: 10.1055/s-0039-1700545. [Epub ahead of print]"
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Factor Xa inhibitor: Patients on treatment with Apixaban, Edoxaban or Rivaroxaban are included into the evaluation study at the outpatient care unit. Patients receive treatment for a specific clinical indication such as non-valvular atrial fibrillation or venous thromboembolism since one week or longer. During the study visit DOAC Dipstick test and liquid-chromatography mass-specrotmery are performed to identify absence or presence of Factor Xa inhibitor in urine.
  "publication Thromb Haemost. 2019 Nov 8. doi: 10.1055/s-0039-1700545. [Epub ahead of print]"
  Interventions: Diagnostic Test: DOAC Dipstick
- Thrombin inhibitor: Patients on treatment with Dabigatran are included included into the evaluation study at the outpatient care unit. Patients receive treatment for a specific clinical indication such as non-valvular atrial fibrillation or venous thromboembolism since one week or longer. During the study visit DOAC Dipstick test and liquid-chromatography mass-specrotmery are performed to identify absence or presence of Thrombin inhibitor in urine.
  "publication Thromb Haemost. 2019 Nov 8. doi: 10.1055/s-0039-1700545. [Epub ahead of print]"
  Interventions: Diagnostic Test: DOAC Dipstick

INTERVENTIONS:
Diagnostic Test: DOAC Dipstick — Patients collect a sample of urine for analysis.
  "publication Thromb Haemost. 2019 Nov 8. doi: 10.1055/s-0039-1700545. [Epub ahead of print]"
  Other Names: test strip for urine analysis"publication Thromb Haemost. 2019 Nov 8. doi: 10.1055/s-0039-1700545. [Epub ahead of print]"

SUMMARY:
This trial is conducted to assess the performance and handling of the in vitro diagnostic (IVD) device for oral direct factor Xa and thrombin inhibitors from urine samples of patients on treatment with direct oral anticoagulants Apixaban, Edoxaban, Rivaroxaban, and Dabigatran (DOAC) in an actual point-of-care (POCT) setting in comparison to results obtained by liquid chromatography tandem mass spectrometry (LC-MS/MS) from urine samples.

This trial is conducted to assess the performance and handling of the IVD for oral direct factor Xa and thrombin inhibitors from urine samples of patients on treatment with DOACs in an actual point-of-care setting in comparison to results obtained by liquid chromatography tandem mass spectrometry (LC-MS/MS) from urine samples.

"publication Thromb Haemost. 2019 Nov 8. doi: 10.1055/s-0039-1700545. [Epub ahead of print]"

DETAILED DESCRIPTION:
This prospective, open-label, controlled, not randomized Performance Assessment will be conducted as a multicenter Performance Assessment in Germany.

The trial investigates the sensitivity and specificity of a POCT for DOAC, i.e., the rate of correct positive, false positive, correct negative and false negative results in the point-of-care setting. The IVD is a test to determine absence or presence of DOAC in urine - Test A tests for oral direct factor Xa inhibitors (rivaroxaban, apixaban, and edoxaban), Test B for oral thrombin inhibitors (dabigatran).

Two groups of patients will be included:

* Test group A: Patients under therapy with oral direct factor Xa inhibitor (rivaroxaban, apixaban, and edoxaban) (n=440)
* Test group B: Patients under therapy with oral thrombin inhibitors (dabigatran) (n=440) No control group of patients not treated with a DOAC is required, as patients take either oral direct factor Xa inhibitors (Test group A) or oral thrombin inhibitors (Test group B), never both. Thus, patients in Test group A are negative for oral thrombin inhibitors and can serve as negative control for Test group B, and vice versa.

The point-of-care test (POCT) is a color-indicator diagnostic medical urine dipstick test for assessing the presence of oral direct factor Xa inhibitor (rivaroxaban, apixaban, and edoxaban) and thrombin inhibitors (dabigatran). The principle of the diagnostic test is based on the development of different colors on the indicator part of the dipstick in the presence or absence of oral direct factor Xa (rivaroxaban, apixaban, and edoxaban) and thrombin inhibitors (dabigatran). The colors for the test were chosen so that they could easily be read by the naked eye, with little possibility of incorrect identification of colors. The results for presence or absence will be compared with the concentration of DOAC analyzed by LC-MS/MS.

Two groups of medications (thrombin inhibitors, factor Xa inhibitors) will be tested with the IVD and test results compared to bioanalytical results in urine.

The objective of the investigation is to show that the proportion of false negative and false positive tests with the IVD is below 5%.

The required sample size to show that the assumed rate of 2.5% false-negative/false-positive tests is statistically significant lower than 5% would require 384 patients per each test group, with α=0.05 and β=0.20 (80% power). Accounting for a potential drop-out rate of 12%, a sample size of n=440 patients per test group was considered adequate to demonstrate adequate performance of the IVD. This sample size has been assessed with the SAS procedure PROC POWER (SAS Institute Inc., Cary, NC, USA, release 9.3) using the ONESAMPLEFREQ statement under the assumption that the test will be conducted as a 1-sided test with a null proportion of 0.05.

For each diagnostic test the proportions of false negative and false positive results will be assessed together with confidence intervals. The urine concentration serves as a gold standard. Furthermore, McNemar tests will be conducted in order to compare the sensitivity, the specificity, accuracy, negative predictive value, positive predictive value and likelihood probability of the two different medications. Kappa coefficients will be calculated in order to quantify the strength of agreement between two diagnostic test methods.

As the study design is not randomized the two groups will be compared according to biographic data (i.e. age, gender, concentration in urine) by common statistical tests (Chi2 test, t-test) in order to investigate their equality. In the case of differences between groups statistical adjustment will be done (i.e. propensity score) in order to avoid the influence of a bias.

The Performance Assessment will be conducted at the patient's family doctor or medical practice/outpatient care unit (referred to as "investigational site" in the following).

The Performance Assessment will consist of a single visit, which is performed during a routine visit at the investigational site.

The Performance Assessment starts with first patient signing informed consent (FPFV) and ends with the last patient providing the last sample (last patient last visit, LPLV).

"publication Thromb Haemost. 2019 Nov 8. doi: 10.1055/s-0039-1700545. [Epub ahead of print]"

ELIGIBILITY:
Inclusion Criteria:

* Fully signed and dated written informed consent
* Age >18 years
* Patient is either under therapy with rivaroxaban, apixaban, and edoxaban or dabigatran for at least 1 week

Exclusion Criteria:

* Patients not able to provide urine samples.
* Patients not able to understand the informed consent or severe mentally disabled.
* Patients in the end-stage of a severe disease.

"publication Thromb Haemost. 2019 Nov 8. doi: 10.1055/s-0039-1700545. [Epub ahead of print]"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on routine treatment with Apixaban, Dabigatran, Edoxaban, and Rivaroxaban since 1 week or longer, an age of >18 years and fulfilling none the exclusion criteria are eligible. The patients participating in this Performance Assessment will be recruited directly at the point of care, i.e., the respective outpatient care unit.
  "publication Thromb Haemost. 2019 Nov 8. doi: 10.1055/s-0039-1700545. [Epub ahead of print]"
Sampling Method: Probability Sample
Enrollment: 880 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Job Harenberg, Professor, Principal Investigator — Pneumonologische Schwerpunktpraxis Heidelberg, Privatpraxis Harenberg
Locations (18):
- Germany (18):
  - Universitätsherzzentrum Bad Krozingen, Klinik für Kardiologie und Angiologie II, Bad Krozingen
  - Herz- und Diabeteszentrum NRW, Klinik für Kardiologie, Bad Oeynhausen
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Gerinnungszentrum Sucker, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Klinikum Coburg GmbH, II. Medizinische Klinik, Coburg
  - Krankenhaus der Augustinerinnen gGmbH, Klinik für Kardiologie und internistische Intensivmedizin, Cologne
  - Klinikum Darmstadt - Gefäßzentrum, Darmstadt
  - Praxis Innere Medizin, Kardiologie und Angiologie, Dessau
  - Städtisches Klinikum Dresden, II. Medizinische Klinik, Dresden
  - Medizinische Fakultät Carl Gustav Carus, Medizinische Klinik und Poliklinik I, Dresden
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Klinik für Kardiologie und Angiologie I, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, II. Medizinische Klinik und Poliklinik, Hamburg
  - Kliniken Landkreis Heidenheim, Heidenheim
  - Zentrum für Blutgerinnungsstörungen, MVZ Labor Dr. Reising-Ackermann und Kollegen, Leipzig
  - Zentrum für Praevention und Rehabilitation, Siegen
  - Die Parkkardiologie, Stahnsdorf

IPD SHARING:
Plan to Share IPD: No
Individual data of patients are collected during the study and stored centrally at DOASENSE GmbH Heidelberg, Germany. They will be shared with other researchers upon request.

REFERENCES:
- [Background] Harenberg J, Du S, Wehling M, Zolfaghari S, Weiss C, Kramer R, Walenga J. Measurement of dabigatran, rivaroxaban and apixaban in samples of plasma, serum and urine, under real life conditions. An international study. Clin Chem Lab Med. 2016 Feb;54(2):275-83. doi: 10.1515/cclm-2015-0389. PMID 26167981
- [Background] Du S, Weiss C, Christina G, Kramer S, Wehling M, Kramer R, Harenberg J. Determination of dabigatran in plasma, serum, and urine samples: comparison of six methods. Clin Chem Lab Med. 2015 Jul;53(8):1237-47. doi: 10.1515/cclm-2014-0991. PMID 25720084
- [Background] Harenberg J, Du S, Kramer S, Weiss C, Kramer R, Wehling M. Patients' serum and urine as easily accessible samples for the measurement of non-vitamin K antagonist oral anticoagulants. Semin Thromb Hemost. 2015 Mar;41(2):228-36. doi: 10.1055/s-0035-1544158. Epub 2015 Feb 15. PMID 25682081
- [Background] Harenberg J, Schreiner R, Hetjens S, Weiss C. Detecting Anti-IIa and Anti-Xa Direct Oral Anticoagulant (DOAC) Agents in Urine using a DOAC Dipstick. Semin Thromb Hemost. 2019 Apr;45(3):275-284. doi: 10.1055/s-0038-1668098. Epub 2018 Aug 22. PMID 30134449
- [Result] Harenberg J, Beyer-Westendorf J, Crowther M, Douxfils J, Elalamy I, Verhamme P, Bauersachs R, Hetjens S, Weiss C; Working Group Members. Accuracy of a Rapid Diagnostic Test for the Presence of Direct Oral Factor Xa or Thrombin Inhibitors in Urine-A Multicenter Trial. Thromb Haemost. 2020 Jan;120(1):132-140. doi: 10.1055/s-0039-1700545. Epub 2019 Nov 8. PMID 31705521
- See also: Homepage DOASENSE GmbH — http://www.doasense.de

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start of study: 18.08.2018 End of study: 10.04.2019 18 centres
Groups:
- Factor Xa Inhibitor: The aim was to include 450 patients on stable treatment with apixaban, edoxaban and rivaroxaban
- Thrombin Inhibitor: The aim was to include 450 patients on stable treatment with dabigatran
Period: Overall Study
Arm/Group | Factor Xa Inhibitor | Thrombin Inhibitor
Started | 467 | 444
Completed | 451 | 429
Not Completed | 16 | 15
Not completed — Protocol Violation | 12 | 12
Not completed — Other | 4 | 3

BASELINE CHARACTERISTICS:
Population: 880 patients with oral intake of a DOAC >7 days patients are included consecutively if inclusion criteria were not meet patients were excluded if patients present an exclusion criteria patients were included comparability of the two patient groups by statistical analysis of baseline demographic data
Groups:
- Factor Xa Inhibitor: Patients on therapy with apixaban, edoxaban and rivaroxaban for at least 7 days
- Thrombin Inhibitor: Patients on therapy with dabigatran for at least 7 days
- Total: Total of all reporting groups
Arm/Group | Factor Xa Inhibitor | Thrombin Inhibitor | Total
Number analyzed (Participants) | 451 | 429 | 880
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 320 | 312 | 632
  >=65 years | 131 | 117 | 248
Age, Continuous [Mean (Full Range); unit: years] | 67 [18 to 93] | 70 [22 to 91] | 68 [18 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 138 | 339
  Male | 250 | 291 | 541
Race/Ethnicity, Customized [Number; unit: participants] | 451 | 429 | 880
Region of Enrollment [Number; unit: participants]
  Germany | 451 | 429 | 880

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Factor Xa and Thrombin Inhibitors Pads of DOAC Dipstick From Urine Samples
Description: Liquid chromatography mass spectrometry versus DOAC Dipstick, qualitative analysis of results
Time Frame: during urine collection and bioanalytical quantification, any time between August 2018 and April 2019
Measure: Mean (95% Confidence Interval); unit: percentage of correct responses
Groups:
- Factor Xa Inhibitor: Patients on treatment with apixaban, edoxaban, rivaroxaban
- Thrombin Inhibitor: Patients treated with dabigatran
Arm/Group | Factor Xa Inhibitor | Thrombin Inhibitor
Number analyzed (Participants) | 451 | 429
percentage of correct responses | 0.973 [0.960 to 0.982] | 0.993 [0.985 to 0.998]
Statistical Analysis 1: Comparison: Factor Xa Inhibitor vs Thrombin Inhibitor; Test type: Non-Inferiority — non-inferiority was chosen; p < 0.05, Chi-squared; Mean Difference (Final Values) = 100, 95% CI 2-sided [90 to 100]; Fisher's exact test

ADVERSE EVENTS:
Time Frame: 2 hours
Description: Adverse Events were not routinely assessed
Groups:
- Factor Xa Inhibitor: Patients on treatment with apxiban, edoxaban and rivaroxaban
- Thrombin Inhibitor: Patients on treatment with dabigatran
Arm/Group | Factor Xa Inhibitor | Thrombin Inhibitor
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT03182829/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT03182829/SAP_001.pdf